CLINICAL TRIAL: NCT05693090
Title: Phase 1 Study of Tipifarnib and Osimertinib in EGFR-mutated Non-Small Cell Lung Cancer
Brief Title: Tipifarnib and Osimertinib in EGFR-mutated Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was withdrawn due to a strategic business decision; no patients were enrolled.
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KO-TIP-015
Expanded Access: NCT04809233 (Available)
Record Dates: First submitted 2022-12-12; First posted 2023-01-20 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: NSCLC
Keywords: EGFR; Tipifarnib; Osimertinib; NSCLC locally advanced; NSCLC metastatic
MeSH Terms: interventions — tipifarnib; osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation Cohort (Experimental): Adult participants with EGFR-mutated Non-Small Cell Lung Cancer
  Interventions: Drug: Tipifarnib; Drug: Osimertinib
- Expansion Cohort (Experimental): Adult participants with EGFR-mutated Non-Small Cell Lung Cancer
  Interventions: Drug: Tipifarnib; Drug: Osimertinib

INTERVENTIONS:
Drug: Tipifarnib — Oral administration
Drug: Osimertinib — Oral administration

SUMMARY:
This is a Phase 1a/b, multicenter, open-label, dose escalation (1a) and dose expansion (1b) study. The purpose of this study is to measure safety, tolerability, and preliminary efficacy with the combination of tipifarnib with osimertinib in patients with advanced/metastatic EGFR-mutated non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing informed consent.
* Histologically or cytologically confirmed stage IIIB (locally-advanced) or IV (metastatic) adenocarcinoma of the lung.
* The tumor harbors an Ex19del or Ex21-L858R substitution (based on tumor tissue or plasma [ctDNA] assessment).
* Treatment-naïve for locally advanced/metastatic EGFR-mutated NSCLC and osimertinib treatment-naïve for NSCLC.
* ECOG performance score of 0 or 1 with no clinically significant deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* Measurable disease by RECIST v1.1 that meets the criteria for selection as a target lesion according to RECIST v1.1.
* Adequate organ function, as evidenced by the laboratory results.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Treatment with any of the following:

  1. Major surgery
  2. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
  3. Medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 (CYP) 3A4 or uridine 5'-diphospho (UDP)-glucuronosyltransferase (UGT), or inhibitors of breast cancer resistance protein (BCRP).
  4. Investigational therapy within 2 weeks of Cycle 1 Day 1
  5. Concurrent and/or other active malignancy that has required systemic treatment within 2 years of first dose of study drug (excluding non-melanoma skin cancer, adjuvant hormonal therapy for breast cancer and hormonal treatment for castration-sensitive prostate cancer)
* Spinal cord compression or symptomatic and unstable brain metastases requiring steroids over the last 4 weeks prior.
* Evidence of severe or uncontrolled systemic diseases.
* Refractory nausea and vomiting, chronic gastrointestinal (GI) diseases, inability to swallow the formulated product, or previous significant bowel resection.
* Clinically significant cardiovascular symptoms or disease.
* Received treatment for unstable angina within prior year, myocardial infarction within the prior 6 months, cerebro-vascular attack within the prior year, history of New York Heart Association grade III or greater congestive heart failure, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
* Past medical history of Interstitial Lung Disease (ILD), drug induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2027-07-27 (Estimated); Study Completion 2027-07-27 (Estimated)

PRIMARY OUTCOMES:
For Dose Escalation determine a safe and tolerable Phase 2 dose of tipifarnib when used in combination with osimertinib | At the end of Cycle 1 (each cycle is 28 days)
  Occurrence of DLTs during first treatment cycle
For Dose Escalation characterize the safety of the combination DLTs will be listed for patients who complete the evaluation period for DLT | DLTs will be evaluated at the end of cycle 1 (28 days), but also through study completion, an average of 1.5 years
  Descriptive statistics of adverse events per NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0)
For Dose Expansion characterize the safety profile of tipifarnib in combination with osimertinib as per NCI CTCAE v5.0 using descriptive statistics of adverse events | Through study completion, an average of 2 years
  Descriptive statistics of adverse events per the NCI CTCAE v5.0
For Dose Expansion characterize the safety profile of tipifarnib in combination with osimertinib as per NCI CTCAE v5.0 using the percentage of patients who discontinue the combination for related adverse events | First 6 cycles of treatment (28 day treatment cycle)
  Percentage of patients who discontinue the combination for tipifarnib and/or osimertinib related adverse events prior to completing 6 cycles of treatment

SECONDARY OUTCOMES:
To evaluate the efficacy of tipifarnib in combination with osimertinib | Assessed every 8 weeks for the first year and every 12 weeks thereafter up to end of study at approximately 2 years
  Objective Response Rate (ORR), measures evaluated according to RECIST v.1.1 assessed by investigator
To evaluate the efficacy of tipifarnib in combination with osimertinib | Assessed every 8 weeks for the first year and every 12 weeks thereafter up to end of study at approximately 2 years
  Duration of Response (DOR) assessed from (CR) or (PR) until (PD), initiation of new anticancer treatment or study withdrawal
To evaluate the efficacy of tipifarnib in combination with osimertinib | Assessed every 8 weeks for the first year and every 12 weeks thereafter up to end of study at approximately 2 years
  Progression-free survival (PFS) measures evaluated according to RECIST v.1.1 assessed by investigator
To study pharmacokinetics (PK) of tipifarnib and osimertinib in combination | Cycles 1-6 (28 day treatment cycle)
  Area under the concentration-time curve (AUC) from time 0 to time of last concentration measured and from time 0 extrapolated to infinity
To study pharmacokinetics (PK) of tipifarnib and osimertinib in combination | Cycles 1-6 (28 day treatment cycle)
  Maximum plasma concentration
To study pharmacokinetics (PK) of tipifarnib and osimertinib in combination | Cycles 1-6 (28 day treatment cycle)
  Time to maximum observed concentration
To study pharmacokinetics (PK) of tipifarnib and osimertinib in combination | Cycles 1-6 (28 day treatment cycle)
  Terminal elimination rate constant
To study pharmacokinetics (PK) of tipifarnib and osimertinib in combination | Cycles 1-6 (28 day treatment cycle)
  Terminal half-life
To study pharmacokinetics (PK) of tipifarnib and osimertinib in combination | Cycles 1-6 (28 day treatment cycle)
  Apparent clearance and apparent volume of distribution
To evaluate circulating tumor DNA (ctDNA) as an indicator or response in both ctDNA positive and negative patients by changes in genetic alterations | Monthly for duration of trial participation (an average of 2 years)
  Determine prevalence of tumor-derived genetic alterations of ctDNA collected at baseline, on-treatment and at disease progression
To evaluate circulating tumor DNA (ctDNA) clearance rates for patients positive at baseline | Monthly for duration of trial participation (an average of 2 years)
  Clearance rates for patients who are ctDNA positive at baseline
To evaluate circulating tumor DNA (ctDNA) time to detection changes associated with disease progression | Monthly for duration of trial participation (an average of 2 years)
  Time to detection of ctDNA changes associated with disease progression

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Providence Medical Group, Santa Rosa, California
  - The Valley Hospital, Ridgewood, New Jersey

IPD SHARING:
Plan to Share IPD: No